CLINICAL TRIAL: NCT00635570
Title: Acceptability of the NuvaRing Among College and Graduate Students
Brief Title: Acceptability of the NuvaRing Among Students
Acronym: ACCEPT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Organon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 14067B; NCT00145899 (obsolete NCT alias)
Record Dates: First submitted 2008-03-05; First posted 2008-03-13 (Estimated); Results first posted 2012-11-07 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2013-06

CONDITIONS: Birth Control Compliance
Keywords: Contraception, Compliance, Acceptability
MeSH Terms: conditions — Patient Compliance | interventions — Moxifloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Contraceptive vaginal ring (Active Comparator): Contraceptive vaginal ring (NuvaRing)
  Interventions: Device: NuvaRing
- Oral contraceptive pill (Active Comparator): Oral contraceptive pill (Ortho Tri-cyclen Lo)
  Interventions: Drug: Ortho Tri-cyclen Lo

INTERVENTIONS:
Drug: Ortho Tri-cyclen Lo — Low dose oral contraceptive
  Arms: Oral contraceptive pill
Device: NuvaRing — Contraceptive vaginal ring
  Arms: Contraceptive vaginal ring

SUMMARY:
The ACCEPT study is a Phase IV trial in which women are randomized to either the NuvaRing® vaginal contraceptive ring or a low dose oral contraceptive to assess compliance, side effects, overall acceptability and intent to continue use of the method. The study is focused on the acceptability of the vaginal ring among female undergraduate or graduate students.

DETAILED DESCRIPTION:
For many women, college is a time of great change that affects one's social and behavioral practices, including sexual behavior. The first part of the NuvaRing ® Acceptability study is an online survey, developed in conjunction with the University of Illinois's Survey Research Laboratory, which examines women's attitudes and beliefs regarding various methods of birth control. The second part of the study is a comparison trial in which the women are randomized to either the NuvaRing ® vaginal contraceptive ring or a low dose oral contraceptive. The women are followed for three months to assess compliance, side effects, overall acceptability and intent to continue use of the method. Ultimately, we would like college women to be well informed about various methods of contraception available to them and to choose the contraceptive method that best suits their lifestyle.

ELIGIBILITY:
Inclusion Criteria:

* over 18
* student enrolled in college or graduate program
* Not have used the contraceptive patch or oral contraceptives within the last month
* Never have used a contraceptive vaginal ring
* Interested in using hormonal contraceptives, specifically NuvaRing and oral contraceptive pills for next 3 months
* In general good health
* Premenopausal with the ability to menstruate

Exclusion Criteria:

* Known or suspected pregnancy
* Pregnancy within 2 months of trial medication
* Past use of any contraceptive vaginal ring
* Hypersensitivity or allergy to NuvaRing or Oral Contraceptives
* Use of investigational drug within 2 months of start of trial medication
* Use of the contraceptive patch or oral contraceptives within past month
* Use of any injectable contraception within 6 months of trial medication
* Planning pregnancy in next 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2008-07; Primary Completion 2009-01 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa L Gilliam, MD, MPH, Principal Investigator — University of Chicago, Section of Family Planning
Locations (3):
- United States (3):
  - University of Chicago, Section of Family Planning, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois

REFERENCES:
- [Background] Gilliam M, Holmquist S, Berlin A. Factors associated with willingness to use the contraceptive vaginal ring. Contraception. 2007 Jul;76(1):30-4. doi: 10.1016/j.contraception.2007.03.009. Epub 2007 May 24. PMID 17586133
- [Derived] Gilliam ML, Neustadt A, Kozloski M, Mistretta S, Tilmon S, Godfrey E. Adherence and acceptability of the contraceptive ring compared with the pill among students: a randomized controlled trial. Obstet Gynecol. 2010 Mar;115(3):503-510. doi: 10.1097/AOG.0b013e3181cf45dc. PMID 20177280

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited 276 participants between March 2006 and December 2008 at two Midwest university-based sites through passive (online and subway advertisements) and active recruitment (referrals from local clinics and health care providers).
Pre-assignment Details: We screened 276 participants, of whom 273 were eligible because 3 of them did not meet inclusion criteria.
Period: Overall Study
Arm/Group | Contraceptive Vaginal Ring | Oral Contraceptive Pill
Started | 136 | 137
Completed | 121 | 126
Not Completed | 15 | 11
Not completed — Lost to Follow-up | 8 | 8
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Did not complete survey | 2 | 1
Not completed — Early termination(No sexual activity) | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Contraceptive Vaginal Ring | Oral Contraceptive Pill | Total
Number analyzed (Participants) | 136 | 137 | 273
Age, Continuous [Mean (Full Range); unit: years] | 22.3 [18 to 38] | 22 [18 to 34] | 22.1 [18 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136 | 137 | 273
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 24 | 20 | 44
  Non-Hispanic White | 66 | 59 | 125
  Non-Hispanic African American | 23 | 28 | 51
  Non-Hispanic Asian | 13 | 15 | 28
  Non-Hispanic other/multiple | 10 | 14 | 24
  Missing | 0 | 1 | 1
Living arrangement [Number; unit: participants]
  Alone | 35 | 32 | 67
  With partner | 16 | 11 | 27
  With others, not partner | 54 | 63 | 117
  With family | 30 | 31 | 61
  Missing | 1 | 0 | 1
Location [Number; unit: participants]
  Dorm | 29 | 34 | 63
  Off campus | 106 | 103 | 209
  Missing | 1 | 0 | 1
Religious preference [Number; unit: participants]
  Catholic | 33 | 36 | 69
  Protestant | 19 | 22 | 41
  Baptist | 11 | 13 | 24
  Other | 18 | 27 | 45
  None | 54 | 37 | 91
  Missing | 1 | 2 | 3
Relationship status [Number; unit: participants]
  Living with a partner in a committed relationship | 19 | 15 | 34
  A committed relationship, not living w/ a partner | 60 | 79 | 139
  Not in a committed relationship | 57 | 41 | 98
  Missing | 0 | 2 | 2
Age at sexual debut [Median (Full Range); unit: Years] — Only of those who had ever had vaginal sexual intercourse ; 125 for contraceptive vaginal ring and 127 for oral contraceptive.
  Years | 17.4 [15 to 26] | 17.8 [13 to 27] | 17.6 [13 to 27]
Vaginal sex in the past month [Number; unit: participants] — Only of those who had ever had vaginal sexual intercourse ; 125 for contraceptive vaginal ring and 127 for oral contraceptive.
  participants
    Yes | 100 | 102 | 202
    No | 25 | 25 | 50
Frequency of sex in current or most recent relationship [Number; unit: participants] — Only of those who had ever had vaginal sexual intercourse ; 125 for contraceptive vaginal ring and 127 for oral contraceptive.
  participants
    None | 4 | 2 | 6
    Once a month or less | 15 | 11 | 26
    2 or 3 times a month | 19 | 18 | 37
    Approximately once a week | 25 | 21 | 46
    2 or 3 times a week | 28 | 37 | 65
    More than 3 times a week | 34 | 36 | 70
    Missing | 0 | 2 | 2
Pregnant ever [Number; unit: participants] — Only of those who had ever had vaginal sexual intercourse ; 125 for contraceptive vaginal ring and 127 for oral contraceptive.
  participants
    Yes | 24 | 12 | 36
    No | 101 | 115 | 216

OUTCOME MEASURES:

1. Primary Outcome: Adherence Rate (Rate of Perfect Method Use)
Description: "Perfect use" was defined as reporting never missing a pill or never removing the contraceptive vaginal ring for more than 2 hours during days 1-21 of all three monthly cycles
Time Frame: For the first 3 months
Measure: Number; unit: Percentage of Participants
Arm/Group | Contraceptive Vaginal Ring | Oral Contraceptive Pill
Number analyzed (Participants) | 136 | 137
Percentage of Participants | 57 | 45
Statistical Analysis 1: Comparison: Contraceptive Vaginal Ring vs Oral Contraceptive Pill; The trial sample size of 300 participants total (150 participants each group) was based on two-sided 5% significance testing with 80% power to detect a difference of 10% in adherence between students in the contraceptive vaginal ring group and oral contraceptive pill group; Test type: Superiority or Other; p = 0.05, Chi-squared, Corrected; Yates's chi-squared test with 1 degree of freedom was used for analysis

2. Secondary Outcome: Satisfaction Rate
Time Frame: at 3 months
Population: 26 participants, 15 out of the contraceptive vaginal ring group and 11 out of the oral contraceptive pill group were excluded. (See the participant flow chart)
Measure: Number; unit: Percentage of Participants
Arm/Group | Contraceptive Vaginal Ring | Oral Contraceptive Pill
Number analyzed (Participants) | 121 | 126
Percentage of Participants
  Satisfaction - Yes | 68 | 71
  Satisfaction - No | 23 | 25
  Missing | 9 | 4
Statistical Analysis 1: Comparison: Contraceptive Vaginal Ring vs Oral Contraceptive Pill; Test type: Superiority or Other; p > 0.05, Chi-squared, Corrected

3. Secondary Outcome: Continuation Rate
Description: Rate of intention to continue the contraceptive method at 3 months
Time Frame: at 3 months
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Contraceptive Vaginal Ring | Oral Contraceptive Pill
Number analyzed (Participants) | 121 | 126
Percentage of Participants
  Continuation - Yes | 43 | 52
  Continuation - No | 52 | 48
  Missing | 5 | 0
Statistical Analysis 1: Comparison: Contraceptive Vaginal Ring vs Oral Contraceptive Pill; Test type: Superiority or Other; p > 0.05, Chi-squared, Corrected

4. Post Hoc Outcome: Continuation Rate
Description: Rate of intention to continue the contraceptive method at 6 months
Time Frame: at 6 month (3 month after the end of the study period)
Population: At 6 months, four from the contraceptive vaginal ring group and three from the oral contraceptive pill group did not complete the 6-month survey and thus were excluded from analysis.
Measure: Number; unit: Percentage of Participants
Arm/Group | Contraceptive Vaginal Ring | Oral Contraceptive Pill
Number analyzed (Participants) | 117 | 123
Percentage of Participants
  Continuation - Yes | 26 | 29
  Continuation - No | 72 | 68
  Missing | 2 | 2
Statistical Analysis 1: Comparison: Contraceptive Vaginal Ring vs Oral Contraceptive Pill; Test type: Superiority or Other; p > 0.05, Chi-squared, Corrected

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Contraceptive Vaginal Ring | Oral Contraceptive Pill
Serious Adverse Events (participants affected / at risk) | 0/136 | 0/137
Other Adverse Events (participants affected / at risk) | 100/136 | 105/137
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Contraceptive Vaginal Ring (N=136) | Oral Contraceptive Pill (N=137)
Bloating (Gastrointestinal disorders) | 73 | 78
Nausea (Gastrointestinal disorders) | 83 | 69
Weight gain (Investigations) | 16 | 18
Headaches (Nervous system disorders) | 93 | 102
Breast swelling (Reproductive system and breast disorders) | 71 | 82
Irregular menstruation (Reproductive system and breast disorders) | 14 | 11
Vaginal discomfort (Reproductive system and breast disorders) | 75 | 58
Vaginal discharge (Reproductive system and breast disorders) | 46 | 15

LIMITATIONS AND CAVEATS:
This study is an randomized controlled trial offering internal but not necessarily external validity. Thus, we do not know whether these findings would be replicable in other populations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes